CLINICAL TRIAL: NCT06905496
Title: Comparison of Outcomes of High Dose Verses Low Dose Caffeine Citrate in the Treatment of Apnea of Prematurity
Brief Title: Apnea of Prematurity Results in Respiratory Distress and Cyanosis. Caffeine Citrate Can Treat It.
Acronym: AOP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Fatima Zahra, Post Graduate Resident, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDLDCC2025; Nishtar Hospital Multan (Other: Nishtar Hospital Multan)
Record Dates: First submitted 2025-03-01; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Apnea of Prematurity
Keywords: caffeine citrate; apnea; prematurity
MeSH Terms: conditions — Apnea; Premature Birth | interventions — caffeine citrate; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Dose Group (Experimental): High dose group will be administered a loading dose of oral caffeine citrate at 40 mg/kg/day followed by a maintenance dose of 20 mg/kg/day for 7 days
  Interventions: Drug: High-Dose; Drug: Low Dose
- Low-Dose Group (Experimental): Low-dose group will receive a loading dose of 20 mg/kg/day and a maintenance dose of 10 mg/kg/day for 7 days
  Interventions: Drug: High-Dose; Drug: Low Dose

INTERVENTIONS:
Drug: High-Dose — Caffeine
  Other Names: Caffeine Citrate 40mg/kg/day
Drug: Low Dose — Caffeine citrate is a combination of caffeine and citric acid, commonly used as a central nervous system stimulant. It is primarily used to treat apnea of prematurity in neonates.

SUMMARY:
High-dose caffeine citrate is more effective than low-dose caffeine citrate in the treatment of apnea of prematurity (AOP). The high-dose group showed fewer apnea episodes, higher extubation success rate, lower extubation failure rate and shorter duration of oxygen therapy

DETAILED DESCRIPTION:
Apnea of prematurity (AOP) is a common condition in preterm infants due to immature respiratory control, affecting up to 80% of those under 1000 grams. It can lead to serious complications, including respiratory distress, pulmonary hemorrhage, and developmental delays. Caffeine citrate, a methylxanthine, is widely used for AOP treatment due to its longer half-life and better absorption compared to theophylline. However, the optimal dosage remains uncertain, with varying practices globally.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a gestational age of ≥32 and <37 weeks at birth on LMP.

  * Diagnosis of apnea of prematurity (AOP) established as per operational definition within the first 10 days of life.
  * Either male or female patients

Exclusion Criteria:

* • Patients diagnosed with Hydrops fetalis (evaluated through medical record).

  * Patients presenting with major congenital or chromosomal anomalies such as anencephaly, spina bifida, congenital heart defects (e.g., tetralogy of Fallot, transposition of the great arteries), or chromosomal disorders (e.g., trisomy 18, Turner syndrome).
  * Presence of a confirmed sepsis through blood culture.
  * Presence of a significant underlying neurological disorder evaluated by history and medical records that could contribute to apnea (e.g., intraventricular hemorrhage with posthemorrhagic hydrocephalus, hypoxic-ischemic encephalopathy)
  * Patients who have been previously treated with caffeine or other methylxanthines for apnea.

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Enhanced Respiratory Stimulation, Effect of Caffeine Citrate on the stimulation of respiratory system of premature individuals | 2-3 days after starting the intervention
  High dose vs low dose caffeine citrate effect in apnea of prematurity. The concentration of caffeine citrate as 40mg high dose and 20mg low dose will be considered. The measurement tool will be percentage of patients recovering from this high vs low concentration.
  The effect of caffeine citrate doses on respiratory stimulation of premature babies will be studied. High doses are expected to improve respiratory distress associated with prematurity. Patients will be clinically assessed after the given doses of caffeine citrate and any improvement, if present, will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Zahra, FCPS, Study Chair — Nishtar Medical University
Locations (1):
- Nishtar Medical Hospital, Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient privacy will be our priority. Consent will be taken from patient for participation in study.